CLINICAL TRIAL: NCT03711604
Title: An Open Label, Compassionate Use Study of Tenalisib (RP6530) in Patients Currently Receiving Treatment on Tenalisib Trials in Hematological Malignancies
Brief Title: Compassionate Use Study of Tenalisib (RP6530)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-1803
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Hematological Malignancies
Keywords: Hematological Malignancies; Tenalisib; RP6530; Compassionate Use
MeSH Terms: conditions — Hematologic Neoplasms | interventions — tenalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tenalisib (Experimental): Participants receive Tenalisib (RP6530) BID Orally
  Interventions: Drug: Tenalisib

INTERVENTIONS:
Drug: Tenalisib — BID Orally
  Other Names: RP6530

SUMMARY:
Tenalisib has been evaluated as an investigational new drug in number of early clinical studies in patients with relapsed/refractory hematological malignancies and demonstrated acceptable safety and promising efficacy in these patients. Since these advanced relapsed/refractory patients have limited therapeutic options, it is reasonable to continue Tenalisib in responding patients post completion of their participation in previous clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be currently receiving treatment with Tenalisib on a previously approved protocol.
2. Patients must have had at least one efficacy evaluation in previous study and should have achieved either SD, PR or CR.
3. Patients must have completed at least 6 cycles of Tenalisib in previous study
4. Ability to swallow and retain oral medication.
5. Female patients of child-bearing potential must consent to use two medically acceptable methods of contraception.
6. Male patients must be willing to use adequate contraceptive measures
7. Willingness and ability to comply with trial and follow-up procedures.
8. Willingness to provide new written informed consent.

Exclusion Criteria:

1. Patient has been discontinued from their previous Tenalisib study 4 weeks prior to entering the compassionate use trial.
2. Patient progressed while receiving Tenalisib therapy in his/her previous study.
3. Pregnant or lactating woman.
4. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.
5. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - University of California, Hellen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Division of Hematology, University of Colorado,, Denver, Colorado
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Georgia (2):
  - Ltd. M.Zodelava Hematology Centre, Tbilisi
  - Medivest - Institute of Hematology and Transfusiology, Tbilisi
- Silesian Healthy Blood Clinic Grosicki, Grosicka Sp.J., Chorzów, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenalisib (RP6530): Participants receive Tenalisib (RP6530) BID orally.
Period: Overall Study
Arm/Group | Tenalisib (RP6530)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Overall, 17 patients were enrolled in this study.
Arm/Group | Tenalisib (RP6530)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.82 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 01
  Native Hawaiian or Other Pacific Islander | 00
  Black or African American | 02
  White | 14
  More than one race | 00
  Unknown or Not Reported | 00

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Adverse Events
Description: To evaluate the safety and tolerability of Tenalisib as single agent. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: 2 years
Population: A total of 17 patients received at least one dose of Tenalisib.
Measure: Count of Participants; unit: Participants
Groups:
- Tenalisib (RP6530): Participants receive Tenalisib (RP6530) orally. Tenalisib (RP6530)
Arm/Group | Tenalisib (RP6530)
Number analyzed (Participants) | 17
Participants | 4

2. Primary Outcome: Time to Disease Progression
Description: Number of patients with a time to progression. The time to progression is calculated from the day of enrollment in the study to disease progression or death due to any cause.
Time Frame: 2 years
Population: A total of 17 patients received at least one dose of Tenalisib.
Measure: Median (Full Range); unit: Months
Arm/Group | Tenalisib (RP6530)
Number analyzed (Participants) | 17
Months | 8.4 [2.77 to 24.01]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. This includes AE, SAE and adverse event of special interest.
Arm/Group | Tenalisib (RP6530)
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib (RP6530) (N=17)
Seizure (Nervous system disorders) | 1 (1)
Hemorrhage intracranial (Nervous system disorders) | 1 (1)
Covid-19 (Infections and infestations) | 2 (3)
Renal Cell Carcinoma (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenalisib (RP6530) (N=17)
Spinal cord compression (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Elevated Aspartate aminotransferase (Investigations) | 2 (3)
Elevated Blood alkaline phosphotase (Investigations) | 2 (5)
Neutrophile count decreased (Investigations) | 2 (7)
Platelet count decreased (Investigations) | 2 (9)
Elevated Troponin (Investigations) | 1 (1)
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Oedema (General disorders) | 2 (2)
Obstruction (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Covid-19 (Infections and infestations) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Supraventriculat extrasystoles (Cardiac disorders) | 1 (1)
Pnuemonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary purpose of this study is to offer patients, who completed a Rhizen-sponsored clinical study without progression, the opportunity to continue to receive Tenalisib on a compassion basis. Thus, the assessments were done in open-label manner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03711604/Prot_SAP_000.pdf